CLINICAL TRIAL: NCT04004130
Title: Ultrasound Imaging of the Subarachnoidal Space at the Lumbar Region in Preterm and Term Newborn Infants
Brief Title: Ultrasound Imaging of Subarachnoidal Space in Newborn Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Szeged University (Other)
Collaborators: Affidea Magyarország (Unknown)
Responsible Party: Principal Investigator, Judit Mari, assistant lecturer, Szeged University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 207/2018
Record Dates: First submitted 2019-06-27; First posted 2019-07-01 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Ultrasound; Newborn Infant
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Ultrasound imaging — Ultrasound imaging of the lumbar spine/subarachnoidal space

SUMMARY:
Based on the ultrasound measurement of CSF/spinal cord ratio in neonates the investigators plan to define a normal range of CSF volume for 0-7 day old newborns. The investigators hypothise to be able to create an ultrasound measurement index/number to predict unsuccessful neonatalal LPs.

DETAILED DESCRIPTION:
Based on the available literature the success rate of neonatal lumbar puncture (LP) is quite low (some articles reporting as low as 50% (unsuccessful LPs including dry taps and traumatic taps)).

Firstly, the investigators would like to set a normal range of CSF:spine ratio (representing the amount of CSF at the expected level of LP) based on the measurements in neonates of different gestational age and postnatal age with assessing ventricular index (VI) on cranial US.

In the next phase of the study the investigators plan to assess the subarachnoidal space/amount of CSF of those neonates whom need LP performed. The investigators hypothise to be able to create an ultrasound measurement index/number that would be able to predict unsuccessful LPs.

ELIGIBILITY:
Inclusion Criteria: All neonates born at the Obstretrics and Gynecology Department, University of Szeged and all treated neonates at the Neonatal Unit, Pediatric Department, University of Szeged

Exclusion Criteria: Hemidynamical instability, Strict minimal handling (eg Pulmonary Hypertension, MAS etc), Total Body Coooling for HIE (Hypoxic Ischemic Encephalopathy)

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2000 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Normal lumbal CSF index in neonates | From Day 1 to Day 7
  Normal range (amount/ratio) of CSF in neonates, influencing the following factors: gestational age, postnatal age, fluid intake, type of delivery.

CONTACTS AND LOCATIONS:
Locations (1):
- Szeged University, Department of Paediatrics, Szeged, Hungary